CLINICAL TRIAL: NCT03742089
Title: Evaluation of Implant Stability and Audiological Benefit of Oticon Medicals BHX Implant in Children Undergoing Surgery for a Percutaneous Bone Anchored Hearing System
Brief Title: Evaluation of the BHX Implant in Children with a BAHS
Status: Completed | Type: Observational
Sponsor: Oticon Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: C52
Record Dates: First submitted 2018-09-24; First posted 2018-11-15 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Hearing Loss, Conductive
MeSH Terms: conditions — Hearing Loss, Conductive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Treatment: Bone Anchored Hearing Surgery using a BHX implant manufactured by Oticon Medical
  Interventions: Device: Bone Anchored Hearing Surgery

INTERVENTIONS:
Device: Bone Anchored Hearing Surgery — This is a observational study of pediatric patients undergoing bone anchored hearing surgery. The collected will be used to assess the implant stability development of the Ponto BHX implant during up to 24 months after implantation in a pediatric population undergoing BAHS. The study will also monitor the Ponto BHX implant safety and survival throughout the study period.

SUMMARY:
The purpose of this study is to in a proactive manner collect high quality data from pediatric patients who have undergone a bone anchored hearing surgery, using the Ponto BHX implant, in clinical practice. This to further increase the knowledge of bone anchored hearing systems in the pediatric population.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have decided to undergo a Bone Anchored Hearing Surgery and receive a Ponto system.
2. Signed informed consent.
3. Patients between 5 - 16 years of age.
4. Patients eligible for one stage surgery.
5. Patients who have been using Ponto sound processor on a soft band for at least 2 weeks.

Exclusion Criteria:

1. Patients who cannot attend follow up visits.
2. Patients with single side deafness (SSD).
3. In surgeon's opinion, any other disorder and condition that may deem the patient unfit to participate in the study.
4. Patients who receive other implant than the Ponto BHX.

   -

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric population eligible for a bone anchored hearing surgery
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2024-09-22 (Actual)

PRIMARY OUTCOMES:
Implant stability | 6 months post surgery
  Implant stability will be assessed using resonance frequency analysis (RFA). This is a non-invasive technique using a SmartPeg (no 55) introduced into the abutment top. A probe is directed to the SmartPeg measuring the vibrations as a test for the stability of the interface between the fixture and the bone (osseointegration). The measurement renders Implant Stability Quotient (ISQ) 'numerical values from 1 to 100'; the higher the ISQ value, the higher the stability. Two perpendicular measurements will be performed at each site. The highest and lowest ISQ value obtained at each time point aree recorded. The Osstell ISQ instrument and SmartPegs from Osstell (Gothenburg, Sweden) will be used. Difference in mean of ISQ low at 6 months compared to surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- The James Cook University Hospital, Middlesbrough, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided